CLINICAL TRIAL: NCT05245227
Title: A Randomized Controlled Trial of Double Simultaneous Uterotonic Agents (Misoprostol Plus Intravenous Oxytocin) Versus Single Agent Regimen (Intravenous Oxytocin Only) to Prevent Early Postpartum Hemorrhage
Brief Title: Double Simultaneous Uterotonic Agents Versus Single Agent Regimen to Prevent Early Postpartum Hemorrhage
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, James Bernasko, MD, Professor, Clinical Obstetrics, Principal investigator, Stony Brook University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB2021-00142
Record Dates: First submitted 2021-11-18; First posted 2022-02-17 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Postpartum Hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Oxytocin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intravenous Oxytocin only (Active Comparator): Patients will receive standard postpartum Oxytocin IV per protocol
  Interventions: Drug: IV Oxytocin
- Misoprostol plus intravenous Oxytocin (Experimental): Patients will receive standard postpartum Oxytocin IV per protocol and also be given Misoprostol 400 mcg sublingual
  Interventions: Drug: Sublingual Misoprostol; Drug: IV Oxytocin

INTERVENTIONS:
Drug: Sublingual Misoprostol — Misoprostol 400 mcg sublingual
  Arms: Misoprostol plus intravenous Oxytocin
Drug: IV Oxytocin — 40 units IV Oxytocin in 1000 mL normal saline

SUMMARY:
To determine the effectiveness of using two medications simultaneously versus one medication, as is standard of care, in preventing early postpartum hemorrhage.

There have been studies that looked at giving two medications and that there were reduced odds of postpartum hemorrhage.

Specific Aim 1: Determine if double simultaneous uterotonic agent regimen (misoprostol and oxytocin) is superior to single agent (oxytocin only) in reducing postpartum hemorrhage.

Specific Aim 2: Determine any potential side effects of a double simultaneous uterotonic agentregimen (misoprostol and oxytocin) versus a single agent (oxytocin only).

DETAILED DESCRIPTION:
Postpartum hemorrhage (PPH) is the leading cause of maternal morbidity and mortality in the world, accounting for a quarter of all maternal deaths globally. Most cases of PPH can be attributed to uterine atony, failure of the uterus to contract in the immediate postpartum period. Efforts to prevent uterine atony and thereby PPH have focused on active clinical management of the third stage of labor (the period between delivery of the infant and placenta) and the administration of uterotonic agents (medication that induces uterine contraction). Universal standard of care to prevent postpartum hemorrhage, according to the American College of Obstetrics and Gynecologists and World Health Organization includes various dose infusions of oxytocin. Additional uterotonics are given if necessary, according to noted blood loss and uterine tone. The best uterotonic(s), combination, route, and dose, however, remain actively debated. Randomized controlled trials have not proven that misoprostol is superior to oxytocin or methergine to treat postpartum hemorrhage, but it is a medication that is often used conjunctively or after other agents fail. A Cochrane review of treatment of primary postpartum hemorrhage revealed that oxytocin, ergot alkaloids (i.e., methergine), and combined oxytocin-ergot alkaloid administration were equally effective in preventing PPH in the general obstetric population, whereas prostaglandins alone (i.e., misoprostol) were not. In an effort to determine the benefit of a simultaneous double uterotonic agent regimen in the prevention of PPH, the investigators propose to conduct a controlled trial in which women will be randomly assigned to an intervention group (buccal misoprostol and intravenous oxytocin administered simultaneously) versus a control group (standard of care, intravenous oxytocin alone).

ELIGIBILITY:
Inclusion Criteria:

- All women 18 years and older admitted to delivery at Stony Brook University hospital who agree to participate in the study

Exclusion Criteria:

* Women under 18 years old
* Women with known coagulation disorders
* Women with planned cesarean hysterectomy
* Women with known placental accreta spectrum disorders
* Women with known allergy to prostaglandins

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients will be female postpartum patients
Enrollment: 1358 (Estimated)
Dates: Start 2025-01-27 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Determine if double simultaneous uterotonic agent regimen (misoprostol and oxytocin) is superior to single agent (oxytocin only) in changing postpartum hemorrhage blood loss volume. | through study completion, an average of 1 year
  Determine if double simultaneous uterotonic agent regimen (misoprostol and oxytocin) is superior to single agent (oxytocin only) in changing postpartum hemorrhage.

SECONDARY OUTCOMES:
Determine serious adverse outcomes of a double simultaneous uterotonic agent regimen (misoprostol and oxytocin) versus a single agent (oxytocin only) that is documented in the medical record. | through study completion, an average of 1 year
  Determine any potential side effects of a double simultaneous uterotonic agent regimen (misoprostol and oxytocin) versus a single agent (oxytocin only).

CONTACTS AND LOCATIONS:
Locations (1):
- Stony Brook University, Stony Brook, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided